CLINICAL TRIAL: NCT04124731
Title: SUNRISE: A Phase II Randomized Control Study of Sintilimab Combined With Anlotinib Versus Standard Platinum-based Chemotherapy as a First-line Treatment in Patients With Advanced NSCLC
Brief Title: Combination Therapy of Sintilimab and Anlotinib as a First-line Treatment in Advanced NSCLC (SUNRISE)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Professor, Director of Pulmonary Medicine at Shanghai Chest Hospita, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNRISE
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma; Non-small Cell Lung Cancer
Keywords: Advanced; Non-Small Cell Lung Cancer; Sintilimab; PD-1; Anlotinib; Anti-angiogenisis
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; anlotinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab plus anlotinib (Experimental): Sintilimab and anlotinib combination therapy
  Interventions: Drug: sintilimab plus anlotinib
- Control (Active Comparator): Standard platinum-based chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: sintilimab plus anlotinib — Sintilimab 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21
  Arms: Sintilimab plus anlotinib
Drug: Chemotherapy — 1. Pemetrexed combined with platinum regimen (non-squamous cell carcinoma): pemetrexed 500mg/m2, intravenous infusion on the first day of each cycle, cisplatin 75mg/m2 or carboplatin AUC 5, intravenous infusion on the first day of each cycle, 1 cycle every 3 weeks (Q3W), 4 cycles in total. Patients who did not progress after 4 cycles received maintenance monotherapy with pemetrexide at the same dose as before.
  2. Gemcitabine combined with platinum regimen (squamous cell carcinoma): gemcitabine 1250mg/m2, intravenous infusion on day 1 and day 8 of each cycle, cisplatin: 75mg/m2 or carboplatin: AUC 5, intravenous infusion on day 1 of each cycle, 1 cycle every 3 weeks (Q3W), 4-6 cycles in total.
  Arms: Control

SUMMARY:
This is an open label, multi-center, randomized control phase II trial, to compare the efficacy and safety of sintilimab combined with anlotinib versus standard platinum-based chemotherapy as a first-line treatment in advanced NSCLC patients without driven-gene mutations.

DETAILED DESCRIPTION:
This is an open label, multi-center, randomized control study comparing the combination of sintilimab and anlotinib with standard platinum-based chemotherapy in treat-naïve advanced (unresectable stage IIIB, IIIC and IV patients without driven-gene mutations) NSCLC patients. Eligible subjects are 1:1 randomized into the experimental group (sintilimab combined with anlotinib) or the control group (standard platinum-based chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before initiation of any study procedures
2. Age ≥ 18 years and ≤ 75 years
3. Histologically or cytologically confirmed NSCLC, with unresectable local advanced or metastatic disease (stage IIIB-IV according to NSCLC staging version 8)
4. Epidermal Growth Factor Receptor (EGFR)/ Anaplastic Lymphoma Kinase (ALK) wild type non-small cell lung cancer
5. Sufficient qualified tumor tissue or Paraffin-embedded slides are provided to detect the expression of PD-L1 (TPS, 22C3 antibody).
6. At least 1 measurable disease according toRECIST 1.1
7. None previous chemotherapy or targeted therapy. Adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment
8. Expected survival over 3 months
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
10. Brain metastasis patients with no symptoms or stable symptoms after local treatment are eligible, provided they meet all of the following conditions:

1) measurable lesions outside the central nervous system 2) no central nervous system symptoms or no aggravation of symptoms for at least 2 weeks 3) patients who did not require glucocorticoid therapy or who discontinued glucocorticoid therapy within 3 days before the first study drug administration 11. Patients are allowed to receive palliative radiotherapy (including craniocerebral radiotherapy for symptomatic brain metastases) at least 1 week prior to enrollment and return to less than or equal to 1 degree of radiosurgery toxicity (CTCAE 5.0, excluding alopecia).

12. Adequate hematologic and organ function defined by the following laboratory results obtained within 14 days prior to randomization: 13. For female patients of childbearing age, a urine or serum pregnancy test should be administered within 3 days prior to the first study drug administration (day 1 of cycle 1) and results should be negative. If a urine pregnancy test does not confirm a negative result, a blood pregnancy test is required. Non-childbearing female were defined as those who had been postmenopausal for at least 1 year or who had undergone surgical sterilization or hysterectomy.

14. If pregnancy is potential, all patients (male and female) are required to use contraception with an annual failure rate of less than 1% for the entire treatment period up to 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration).

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma); Small cell lung cancer (including small cell cancer and non-small cell mixed lung cancer).
2. Patients with cavernous squamous cell carcinoma or imaging suggesting infiltration/invasion of large blood vessels or other high bleeding risk factors evaluated by the investigators.
3. Active hemoptysis within 2 weeks before first drug administration (at least 1/2 teaspoon blood spilt at one time);
4. Received radiotherapy before administration of the first study drug, which met one of the following conditions:

1) ≥30% of bone marrow had received radiotherapy within 14 days before treatment 2) received radiotherapy for lung lesions within 6 weeks before treatment with >30Gy dose (enrolled subjects must recover from the toxicity of previous radiotherapy to level 1 or below, do not need glucocorticoid treatment and have no history of radiation pneumonia) 3) the end time of palliative radiotherapy should be within 7 days before the first study drug administration 5. Major surgical treatment within 3 weeks of the first study drug administration (except for biopsy surgery) 6. Have Participated in other clinical studies or less than 4 weeks before the end of treatment in the previous clinical study 7. Previously diagnosis as other malignant tumors within 5 years prior to the first dose of study treatment, with the exception of: skin basal cell carcinoma or squamous cell carcinoma with radical treatment, and/or carcinoma in situ underwent radical resection 8. Prior treatment with PD-1 inhibitor, PD-L1 inhibitor, CTLA4 inhibitor, or anti- angiogenic treatment.

9. A history of active autoimmune disease requiring systemic treatment (e.g. using drugs for disease remission, corticosteroids or immunosuppressor) within 2 years prior to the first dose of study treatment. Substitution therapy (e.g. thyroxine, insulin or physiological corticosteroids for treating adrenal or pituitary dysfunction) is not considered as a systemic treatment.

10. Received a traditional Chinese medicine with anti-tumor effect, or an immunomodulatory drug (thymosin, interferon, interleukin) within 2 weeks before the first dose, or received major surgery within 3 weeks before the first dose 11. Systemic steroid therapy or any other form of immunosuppressive therapy performed within 7 days prior to the first dose of study (physiologic dose is allowed).

12. The presence of clinically uncontrollable pleural effusion/peritoneal effusion 13. Have received a physical organ or blood system transplant 14. allergic to the active ingredients or excipients of the drugs studied, such as sintilimab, pemetrexed, gemcitabine, carboplatin, cisplatin, etc.

15. Patients with multiple factors that affect oral medications (such as inability to swallow, gastrointestinal resection, chronic diarrhea, and intestinal obstruction) 16. Patients with bleeding tendencies (such as active gastrointestinal ulcers) or treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; Small doses of warfarin (≤1mg/d), small doses of heparin (≤ 12,000 U/d) or small doses of aspirin (≤100mg/d) are allowed for prophylactic purposes, provided that the international standardized ratio of prothrombin time (INR) ≤1.5 17. Patients with severe arteriovenous thrombosis, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism, which occurred within 6 months before the first treatment 18. Not fully recovered from toxicity and/or complications resulting from any intervention prior to initiation of treatment (i.e., ≤1 or baseline, excluding fatigue or hair loss); 19. A history of human immunodeficiency virus (HIV) infection (ie, HIV 1/2 antibody positive) is known.

20. Untreated active hepatitis B; 21. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection) 22. Vaccination of live vaccine within 30 days before the first dose (1st cycle, 1st day); 23. Pregnant or lactating women 24. Any serious or uncontrolled systemic diseases 25. Any medical history or evidence of disease that may interfere with the outcome of the study, or other conditions that the investigator considers inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Objective Respond Rate (ORR) | up to 24 months after enrollment or study close
  ORR (per RECIST 1.1 as assessed by the investigator) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months after enrollment or study close
  PFS (per RECIST 1.1 as assessed by the investigator) is defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression)
Disease Control Rate (DCR) | up to 24 months after enrollment or study close
  DCR (per RECIST 1.1 as assessed by the investigator) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD).
Duration of Response (DoR) | up to 24 months after enrollment or study close
  DoR (per RECIST 1.1 as assessed by the investigator) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) until the date for the first documented response of progressive disease (PD) or death in the absence of progression.
Overall Survival (OS) | up to 24 months after enrollment or study close
  OS (per RECIST 1.1 as assessed by the investigator) is defined as the time from the date of randomisation until death due to any cause.